CLINICAL TRIAL: NCT06184763
Title: Evolution of the 6-minute Walk Test in Patients Treated With ELEXACAFTOR / TEZACAFTOR / IVACAFTOR
Acronym: TEMETI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 23-5232; Easydore (Other: 69HCL23_1322)
Record Dates: First submitted 2023-12-15; First posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; CFTR modulators; 6-minutes walk test; physical activity
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ELEXACAFTOR/TEZACAFTOR/ IVACAFTOR treated patients: Patients ≥ 12 years old with cystic fibrosis followed at the Renee Sabran Hospital, heterozygous for the F508del mutation of the CFTR gene, treated with ELEXACAFTOR/ TEZACAFTOR/ IVACAFTOR.
  Intervention: 6-minute walk test before and after starting treatment.
  Interventions: Other: 6-minute walk test

INTERVENTIONS:
Other: 6-minute walk test — 6-minute walk test in a 40-metre corridor. Included patients are used to performing this test, which is part of the standard care performed during patient follow-up, at least once a year.
  Parameters collected during the test: distance walked, minimum SpO2, average SpO2, maximum heart rate, average heart rate, average heart rate over the last 2 minutes, dyspnea scale.

SUMMARY:
The aim of the study is to identify a link between the new CFTR modulators and physical activity in cystic fibrosis patients.

The triple combination of CFTR modulators (ELEXACAFTOR / TEZACAFTOR/ IVACAFTOR) has recently changed the management of cystic fibrosis.

This treatment has been shown to rapidly improve patients' respiratory function, with a gain in FEV1 at 1 month ranging from 10.4% to 13.6%. It also reduces the number of respiratory exacerbations and improves the nutritional status and quality of life of treated patients.

To date, there is limited data on the impact of these new therapies on physical activity. Few studies have investigated changes in exercise or physical activity parameters under ELEXACAFTOR / TEZACAFTOR/ IVACAFTOR.

The 6-minute walk test is a validated field test used routinely to assess the exercise capacity of patients with chronic respiratory diseases, including cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 12 years with cystic fibrosis, heterozygous for the F508del mutation of the CFTR gene, treated with ELEXACAFTOR/ TEZACAFTOR/ IVACAFTOR.
* Patients followed in the respiratory diseases department of the Renee Sabran Hospital
* 6-minute walked test performed in the year preceding initiation of ELEXACAFTOR / TEZACAFTOR/ IVACAFTOR
* 6-minute walked test performed after treatment initiation (between the 3rd month and the 14th month)
* No opposition to participation

Exclusion Criteria:

* - Age < 12 years
* Pregnancy
* Discontinuation or reduction in dosage of ELEXACAFTOR/ TEZACAFTOR/ IVACAFTOR
* Patients objecting to the use of their data for research purposes

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cohort: cystic fibrosis patients followed in the respiratory diseases department of the Renee Sabran Hospital (approximately 100 patients)
Sampling Method: Non-Probability Sample
Enrollment: 73 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
distance walked in the 6-minute walk test (metres) | between the 3rd month and the 14th month post treatment initiation
  Distance walked in the 6-minute walk test, compared before and after the introduction of ELEXACAFTOR/ TEZACAFTOR/ IVACAFTOR.

CONTACTS AND LOCATIONS:
Locations (1):
- Respiratory diseases department, Renee Sabran Hospital (Hospices civils de Lyon), Giens, France

IPD SHARING:
Plan to Share IPD: No